CLINICAL TRIAL: NCT03965793
Title: Individualized Fluid and Vasopressor Administration in Surgical Patients: A Randomized Controlled Trial
Brief Title: Individualized Fluid And Vasopressor Administration In Surgical Patients
Acronym: INFIVASP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP190369
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Intraoperative Hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual management of hypotension (Active Comparator): Fluid and vasopressor will be managed as standard practice ( manually infusion of both fluid and vasopressors) following the investigators manual individualized hemodynamic protocol.(objective being to keep both stroke volume and MAP within 90 % of the target values)
  Interventions: Device: Automated management of hypotension
- Automated management of hypotension (Experimental): Fluid and vasopressor will be managed with a novel active clinical decision support system to guide fluid administration and automated closed-loop system to maintain MAP within 90% of patient' baseline.
  Interventions: Device: Automated management of hypotension

INTERVENTIONS:
Device: Automated management of hypotension — Fluid and vasopressor will be administered based on a novel automated clinical decision support system.

SUMMARY:
The purpose of this study is to compare two different strategies of intraoperative mean arterial pressure (MAP) and stroke volume index management in high-risk patients undergoing major abdominal and orthopedic surgery (manual versus automated) The investigators hypothesis is that the automated group will spend less time during surgery in hypotension (defined as a MAP<90% of patient's MAP baseline) compared to the manual group.

DETAILED DESCRIPTION:
The maintenance of MAP is essential for organ perfusion pressure. Intraoperative hypotension is a frequent complication both after induction and during maintenance of anaesthesia, ranging from 5% to 75% depending on the chosen definition. Tissue hypoperfusion exposes to the occurrence of a systemic inflammatory response syndrome and is a key determinant of postoperative complications. Persistent intraoperative hypotension has been reported as an important prognostic factor of postoperative morbidity and mortality. Adequate treatment of arterial hypotension is therefore of particular importance during surgery. However, the avoidance of hypotension includes the infusion of vasopressor and/or fluid to optimize perfusion pressure. The manual adjustment of vasopressor administration has been shown to be suboptimal.

Recently, a paper published in the JAMA journal demonstrated that among patients undergoing high-risk surgery, the maintenance of blood pressure within 10% of patient's baseline systolic blood pressure resulted in less postoperative organ dysfunction compared to standard MAP management.

Today, the investigators have an automated clinical decision support system that help ease the administration of both fluid and vasopressors during surgery (individualized fluid and vasopressor administration). The department of the investigators has recently implemented a manual hemodynamic protocol to optimize fluid and vasopressor. The goal is to maintain stroke volume index within 90% of the optimal stroke volume via mini fluid challenge of crystalloid solution (100 ml) following the French guidelines and to maintain MAP within 90 % of patient's baseline MAP. This protocol has been called : Individualized Fluid and vasopressor protocol (because based on patient's values) The purpose of this study is therefore to compare two different strategies of intraoperative mean arterial pressure (MAP) and stroke volume index management in high-risk surgical patients (manual versus automated and decision support guided) The investigators hypothesis is that automated group will spend less time during surgery in hypotension (defined as a MAP<90% of patient's MAP baseline) compared to the manual group because patient's stroke volume and MAP will be better maintained during surgery (within 10% of patient' targets).The decision support system will remind the clinician when to administer a bolus of fluid to maintain stroke volume index within 10% of the optimize stroke volume index value and an automated closed-lopp system will titrate norepinephrine to keep MAP within 10% of patient's MAP target. The study will thus compare an individualized hemodynamic protocol (already in place in our institution) applied manually to a decision support-and closed-loop guided- individualized hemodynamic protocol (intervention group).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients scheduled for major abdominal and orthopedic surgery equipped with a cardiac output monitoring device.

Exclusion Criteria:

* Patients < 18 years old
* cardiac arrythmia (atrial fibrillation)
* Pregnant woman

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-10-27 (Actual); Primary Completion 2020-07-26 (Actual); Study Completion 2020-07-26 (Actual)

PRIMARY OUTCOMES:
Percentage of surgery time in hypotension | at day 1
  Percentage of surgery time in hypotension (defined as the percentage of case time the patient will spend with a MAP < 10% of patient's MAP Baseline)

SECONDARY OUTCOMES:
Postoperative complications incidence | at DAY 30
  Number of postoperative complications at day 30 post surgery among the 9 items (postoperative nausea and vomiting, delirium, wound infection, urinary infection, pneumonia, acute kidney injury incidence, paralytic ileus, other infections, readmission to hospital within the 30 days post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Joosten, MD PhD, Principal Investigator — Bicetre hospital, APHP.
Locations (1):
- Bicetre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No